Unique Protocol ID: SE 312/2021

Brief Title: Adaptation of Pediatric Speech Audiometry Tests Into Other Languages

Official Title: Methodological Guide for the Adaptation of Pediatric Speech Audiometry

Tests Into Other Languages

25 August 2025

#### Semmelweis University Budapest



## Department of Voice, Speech and Swallowing Therapy

#### **Parental Consent Form and Questionnaire**

#### Introduction

Your child is invited to participate in a research study that aims to adapt and validate a Hungarian version of a pediatric speech audiometry test. This research will help in the development of reliable hearing assessments for children in Hungary.

#### **Procedures**

Your child will be asked to participate in a hearing screening and a speech recognition test using familiar images.

#### **Voluntary Participation**

Participation is entirely voluntary. You may withdraw your child from the study at any time without any consequences.

#### **Risks and Benefits**

There are no anticipated risks related to participation. Participation may benefit future improvements in pediatric hearing assessments in Hungary.

#### Confidentiality

All data will be anonymized and handled confidentially. Your child's name will not appear in any publications or reports.

#### **Contact Information**

For questions or concerns, please contact: Dr. Gergely Vasvári; Semmelweis University; Email: g.vasvari@gmail.com

#### **Parental Consent Statement**

| $\square$ I have read and understood the information above. I volun participation in this study. | tarily consent to my child's |
|---|---|
| participation in this study. | |
| Name of Parent/Guardian: | |
| Signature of Parent/Guardian: | _ |
| Date: / / | |

### Semmelweis University Budapest



# Department of Voice, Speech and Swallowing Therapy

## **Questionnaire for Parents**

| Participant Information |
|---|
| Child's Identifier (or Name): |
| Date of Birth: / / |
| Sex: □ Male □ Female |
| Kindergarten attended: |
| Inclusion Criteria Checklist |
| Please answer the following: |
| 1. Does your child currently have symptoms of an upper respiratory tract infection? $\square$ Yes $\square$ No |
| 2. Has your child been diagnosed with any speech-language developmental disorders? $\Box$<br>Yes $\Box$<br>No |
| 3. Has your child been diagnosed with any cognitive disorders? ☐ Yes ☐ No |
| 4. Does your child have any hearing problems known to you? ☐ Yes ☐ No |
| If you answered Yes to any of the above, please provide additional details (optional): |
| Optional |
| Is your child regularly exposed to other languages at home? $\ \square$ Yes $\ \square$ No |
| If ves. which language(s)? |